CLINICAL TRIAL: NCT02546609
Title: A Randomized, Blinded, Placebo-Controlled Study To Evaluate The Effect Fixed-Dose Leucine, Metformin, Sildenafil Combinations(NS-0200) Versus Placebo On Hepatic Fat Assessed By MRI In Non Alcoholic Fatty Liver Disease Patients
Brief Title: The Effect Of NS-0200 Versus Placebo On Hepatic Fat Content In Patients With Non Alcoholic Fatty Liver Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NuSirt Biopharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NS-0200-01
Record Dates: First submitted 2015-09-03; First posted 2015-09-11 (Estimated); Results first posted 2018-05-02 (Actual); Last update posted 2018-05-02 (Actual); Status verified 2018-04

CONDITIONS: NAFLD
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Leu Met Sil 0.5mg (Experimental): Leu-Met-Sil 0.5: 3 capsules BID consisting of 2 capsules containing 550 mg L-leucine each and 1 capsule containing 500 mg metformin and 0.5 mg of sildenafil.
  Interventions: Drug: Leu-Met-Sil 1.0
- Leu Met Sil 1.0mg (Experimental): Leu-Met-Sil 1.0: 3 capsules BID consisting of 2 capsules containing 550 mg L-leucine each and 1 capsule containing 500 mg metformin and 1.0 mg of sildenafil.
  Interventions: Drug: Leu-Met-Sil 0.5; Drug: Leu-Met-Sil 1.0
- Placebo (Placebo Comparator): Placebo: 3 capsules BID containing 99% Avicel PH302 and 1% magnesium stearate (w/w)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Leu-Met-Sil 0.5 — NS-0200 low dose
  Other Names: NS-0200-0.5
  Arms: Leu Met Sil 1.0mg
Drug: Leu-Met-Sil 1.0 — NS-200 high dose
  Other Names: NS-0200-1.0
  Arms: Leu Met Sil 0.5mg; Leu Met Sil 1.0mg
Drug: Placebo — Placebo
  Other Names: Control arm
  Arms: Placebo

SUMMARY:
The goal of this study is to determine if NS-0200 can reduce the amount of liver fat in patients diagnosed with non-alcoholic fatty liver disease (NAFLD). This study will compare two doses of NS-0200 to placebo in NAFLD patients.

DETAILED DESCRIPTION:
This is a randomized, 16-week, placebo-controlled, double-blind study to evaluate the effect of two fixed-dose combinations of leucine, metformin and sildenafil, NS-0200 compared to placebo, on the reduction of liver fat in patients diagnosed with non-alcoholic fatty liver disease (NAFLD). Subjects meeting all the inclusion criteria and no exclusion criteria will be randomized to one of three study arms.

The primary objective of this study is to evaluate the change in hepatic fat content assessed by proton-density-fat-fraction (PDFF) employing magnetic resonance imaging (MRI) in subjects from : Screening/Visit 2 (Day-7/Week-1) to Study Termination/Visit 8 (Day 112/Week 16) receiving two fixed-dose combinations of leucine, metformin and sildenafil compared to placebo. Secondary objectives will also assess changes in serum alanine aminotransferase (ALT) activity, change in circulating cytokeratin 18, a surrogate marker of necro-inflammation, change in HbA1c, change in fasting glucose, insulin and insulin sensitivity, change in blood lipids such as cholesterol, LDL, HDL, triglycerides, and changes in in C-reactive protein. In addition this study will evaluate the safety and tolerability of NS-0200.

Patients will have two screening visits, the first to determine their eligibility based on lab tests and the second based on the percentage of hepatic fat assessed by MRI imaging. Once qualified, patients will be randomly assigned to either one of the treatment groups or the placebo control group and monitored for a total of 16 weeks. Patients will return to the clinic each month for lab tests, and routine examinations. At the conclusion of the treatment period patients will again undergo an MRI scan to examine the percentage of hepatic fat.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 at study entry.
2. Is male, or female and, if female, meets all of the following criteria:

   1. Not breastfeeding
   2. Post-menopausal or negative serum pregnancy test result (human chorionic gonadotropin, beta subunit [β-hCG]) at Screening /Visit 1 (Day-14/Week-2) (not required for hysterectomized females)
   3. If of childbearing potential (including peri-menopausal women who have had a menstrual period within one year) must practice and be willing to continue to practice appropriate birth control (defined as a method which results in a low failure rate, i.e., less than 1% per year, when used consistently and correctly, such as double barrier methods [male condom with spermicide, with or without cervical cap or diaphragm], implants, injectables, oral contraceptives [must have been using for at least the last 3 months], some intrauterine contraceptive devices, tubal ligation, or in an established relationship with a vasectomized partner) during the entire duration of the study.
3. Has been diagnosed with NAFLD via CT (positive for excess liver fat), ultrasound (positive for excess liver fat), MRI (PDFF showing > 15% liver fat) or via biopsy (showing >33% fat) within the past six months. If diagnosis was between 3 and 6 months prior to Screening, an ultrasound (positive for excess liver fat) is required prior to the Screening /Visit 1 (Day-14/Week-2) MRI.
4. Has liver fat (as measured by PDFF via MRI) greater than 15% at Screening/Visit 2 (Day-7/Week-1)
5. Has had ALT levels >30 U/L for men, >19 U/L for women measured within 8 weeks of enrollment
6. Has an HbA1c equal to or less than 9% at Screening /Visit 1 (Day-14/Week-2)
7. Has a BMI between 25kg/m2 and 40 kg/m2
8. Otherwise stable health for preceding twelve weeks
9. Clinical laboratory tests (hematology, clinical chemistry, and urinalysis) either normal or with abnormalities consistent with NAFLD.
10. Is able to read, understand, and sign the informed consent forms (ICF) and, when applicable, an authorization to use and disclose protected health information form (consistent with Health Insurance Portability and Accountability Act of 1996 [HIPAA] legislation), communicate with the investigator, and understand and comply with protocol requirements.

    -

Exclusion Criteria:

1. Clinically significant renal dysfunction defined as a serum creatinine concentration >1.4 mg/dL (females) or >1.6 mg/dL (males) or a blood urea nitrogen concentration >45 mg/dL at screening.
2. Use of any of the following medications:

   1. Metformin
   2. Combination drugs that include Metformin
   3. Sildenafil
   4. Tadalafil
   5. Vardenafil
   6. Pioglitazone
   7. Rosiglitazone
   8. Short acting insulins
   9. An alpha blocker
   10. Oral nitrates
   11. Medications associated with increased hepatic steatosis
   12. Insulins
   13. OCT2/MATE inhibitors (e.g. cimetidine, quinidine, and pyrimethamine)

       * Methotrexate
       * Tamoxifen
       * Corticosteroids (Nasal steroids are allowed if the subject has been on a stable dose for the past 12 weeks and the dose employed does not exceed the maximal recommended dose.)
       * Estrogens
       * Amiodarone
       * Valproic acid
       * Coumadin
       * Isoniazide
       * Nucleoside analogues used for the treatment of HIV infections
   14. Any dietary supplement other than multi-vitamins
3. Evidence of significant alcohol consumption (defined as >7 drinks/week for females and >14 drinks/week for males) within 6 months prior to randomization or presence or suspicion of other forms of chronic liver disease (e.g., cirrhosis, autoimmune hepatitis (>1:160 ANA), Wilson's disease, Hemochromatosis (Ferritin >1000 ug/L and percent iron saturation >45%), hepatitis A, B or C)
4. Has a clinically significant medical condition that could potentially affect study participation and/or personal well-being, as judged by the investigator, including but not limited to the following conditions:

   1. Unable to undergo MRI or contraindications for MRI procedure
   2. History of cardio- or cerebro-vascular disease event within the previous 6 months
   3. Requires anti-coagulation therapy
   4. Gastrointestinal disorders including, but not limited to, the following: pancreatitis, inflammatory bowel disease, or other diseases associated with malabsorption or persistent abdominal discomfort
   5. Endocrine disorders other than type 2 diabetes and hypothyroidism on stable replacement therapy
   6. Chronic infection (e.g., tuberculosis, human immunodeficiency virus infection, hepatitis A virus, hepatitis B virus, or hepatitis C virus)
   7. Neurological or psychiatric diseases that preclude valid execution of informed consent or may interfere with the subject's compliance with study procedures (e.g., major depressive disorder within the last 2 years, a history of suicidal behavior in the last 3 months)
   8. History of other psychiatric disorders including schizophrenia and bipolar disorder)
5. Participation in a weight loss program within the past 3 months.
6. Weight change ≥5% during the past month.
7. History of substance abuse (including alcohol abuse as defined above) in the past 3 months or a positive screen for drugs of abuse or alcohol at screening.
8. Has received any investigational drug within 3 months of Screening.
9. Has donated blood within 3 months before Screening or is planning to donate blood during the study.
10. Has had a serious infection, such as pneumonia in the previous 12 weeks
11. Has known allergies or hypersensitivity to metformin, sildenafil or leucine
12. Is an immediate family member (spouse, parent, child, or sibling; biological or legally adopted) of personnel directly affiliated with the study at the clinical study site, or NuSirt Biopharma.
13. Is employed by NuSirt Biopharma (defined as an employee, temporary contract worker, or designee responsible for the conduct of the study).

    -

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2015-11-19; Primary Completion 2016-11-30 (Actual); Study Completion 2017-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Orville Kolterman, MD, Study Director — NuSirt Biopharma
Locations (13):
- United States (13):
  - Catalina Research Institute, Chino, California
  - University of California San Diego, San Diego, California
  - Rocky Mountain Research, Wheat Ridge, Colorado
  - Atlanta Gastroenterology Associates, Atlanta, Georgia
  - GI Specialists of Georgia, Marietta, Georgia
  - Northwestern University, Chicago, Illinois
  - Indiana University, Indianapolis, Indiana
  - University of North Carolina Chapel Hill, Chapel Hill, North Carolina
  - Sterling Research, Cincinnati, Ohio
  - Premier Clinical Research, Clarksville, Tennessee
  - Gastro One, Germantown, Tennessee
  - Quality Medical Research, Nashville, Tennessee
  - Virginia Commonwealth University, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nedrud MA, Chaudhry M, Middleton MS, Moylan CA, Lerebours R, Luo S, Farjat A, Guy C, Loomba R, Abdelmalek MF, Sirlin CB, Bashir MR. MRI Quantification of Placebo Effect in Nonalcoholic Steatohepatitis Clinical Trials. Radiology. 2023 Mar;306(3):e220743. doi: 10.1148/radiol.220743. Epub 2022 Nov 1. PMID 36318027
- [Derived] Zemel MB, Kolterman O, Rinella M, Vuppalanchi R, Flores O, Barritt AS 4th, Siddiqui M, Chalasani N. Randomized Controlled Trial of a Leucine-Metformin-Sildenafil Combination (NS-0200) on Weight and Metabolic Parameters. Obesity (Silver Spring). 2019 Jan;27(1):59-67. doi: 10.1002/oby.22346. PMID 30569637

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects meeting all inclusion criteria and no exclusion criteria were randomized to one of the three treatment arms in the ratio of 1:1:1. Adult males and females (age 18-75) with CT, MRI, biopsy, or ultrasound consistent with NAFLD within the past 6 months.
Groups:
- Placebo: 3 capsules BID containing 99% Avicel PH302 and 1% magnesium stearate (w/w)
  Placebo: Placebo
- Leu Met Sil 0.5mg: 3 capsules BID consisting of 2 capsules containing 550 mg L-leucine each and 1 capsule containing 500 mg metformin and 0.5 mg of sildenafil.
  Metformin: 500 mg Metformin BID
  Leucine: 1100 mg Leucine BID
  Sildenafil Citrate 0.5 mg: Sildenafil 0.5 mg BID
- Leu Met Sil 1.0mg: 3 capsules BID consisting of 2 capsules containing 550 mg L-leucine each and 1 capsule containing 500 mg metformin and 1.0 mg of sildenafil.
  Sildenafil 1.0 mg: Sildenafil 1.0 mg
  Metformin: 500 mg Metformin BID
  Leucine: 1100 mg Leucine BID
Period: Overall Study
Arm/Group | Placebo | Leu Met Sil 0.5mg | Leu Met Sil 1.0mg
Started | 24 | 35 | 32
Completed | 22 | 24 | 25
Not Completed | 2 | 11 | 7
Not completed — Withdrawal by Subject | 0 | 1 | 2
Not completed — Adverse Event | 0 | 6 | 1
Not completed — Protocol Violation | 0 | 1 | 1
Not completed — Lost to Follow-up | 2 | 3 | 1
Not completed — travel or work schedule restriction | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: Demographic and other baseline characteristics were analyzed using the ITT Population with subjects who met the inclusion criteria.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Leu Met Sil 0.5mg | Leu Met Sil 1.0mg | Total
Number analyzed (Participants) | 24 | 34 | 32 | 90
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 24 | 34 | 27 | 85
  >=65 years | 0 | 0 | 5 | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.3 (10.42) | 45.1 (11.72) | 45.9 (12.71) | 45.7 (11.64)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 21 | 17 | 50
  Male | 12 | 13 | 15 | 40
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 12 | 12 | 30
  Not Hispanic or Latino | 18 | 22 | 20 | 60
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 1
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 1 | 0 | 3
  White | 21 | 31 | 29 | 81
  More than one race | 1 | 1 | 0 | 2
  Unknown or Not Reported | 0 | 1 | 2 | 3
Weight [Mean (Standard Deviation); unit: kg] | 96.83 (15.061) | 94.44 (16.332) | 94.11 (17.225) | 94.96 (16.192)
Height [Mean (Standard Deviation); unit: cm] | 170.1 (9.48) | 169.6 (10.58) | 167 (10.75) | 168.8 (10.34)
Body mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 33.5 (4.534) | 32.60 (3.486) | 33.52 (4.167) | 33.17 (4.008)
Fasting Plasma Glucose [Mean (Standard Deviation); unit: mg/dL] | 108.2 (16.53) | 104.3 (14.28) | 115.4 (27.61) | 109.3 (20.86)
HbA1c [Mean (Standard Deviation); unit: percentage of glycosylated hemoglobin] | 5.59 (0.495) | 5.65 (0.528) | 5.86 (0.738) | 5.71 (0.609)
Childbearing Potential [Count of Participants; unit: Participants] — Population: Childbearing potential is only applicable to the female participants hence the difference in overall population and number analyzed for this category.
  Participants
    number analyzed (Participants) | 12 | 21 | 17 | 50
    Child-bearing potential with adequate birth contro | 3 | 6 | 3 | 12
    Postmenopausal | 1 | 4 | 3 | 8
    Surgically Sterile | 8 | 11 | 11 | 30

OUTCOME MEASURES:

1. Primary Outcome: Change in Hepatic Fat
Description: To evaluate the change in hepatic fat content assessed by proton-density-fat-fraction (PDFF) employing magnetic resonance imaging (MRI).
Time Frame: Baseline, Day 112
Population: For the Per-Protocol Population (N=70), the mean percent change (SD) in hepatic fat content (%) from Baseline to Week 16 (Day 112) for each treatment group was assessed.
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Placebo | Leu Met Sil 0.5mg | Leu Met Sil 1.0mg
Number analyzed (Participants) | 22 | 24 | 24
percentage | -10.046 (17.5335) | 3.083 (25.5230) | -4.013 (24.6302)
Statistical Analysis 1: Comparison: Placebo vs Leu Met Sil 0.5mg; Analysis of variance (ANOVA) model: with treatment group as the factor. Placebo is used as the reference group; Test type: Other; p = 0.0572, ANCOVA
Statistical Analysis 2: Comparison: Placebo vs Leu Met Sil 1.0mg; Analysis of variance (ANOVA) model: with treatment group as the factor. Placebo is used as the reference group; Test type: Other; p = 0.3770, ANCOVA

2. Secondary Outcome: Change in Serum AlanineAaminotransferase (ALT) Levels
Description: Serum AlanineAminotransferase (ALT) will be examined through standard blood chemistry
Time Frame: Baseline, Day 112
Population: For the Per-Protocol Population (N=70), the mean change (SD) in serum ALT levels from Baseline to Week 16 was assessed
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Placebo | Leu Met Sil 0.5mg | Leu Met Sil 1.0mg
Number analyzed (Participants) | 22 | 24 | 24
U/L | -4.1 (20.09) | 1.8 (22.67) | -2.7 (22.96)
Statistical Analysis 1: Comparison: Placebo vs Leu Met Sil 0.5mg; MMRM model: with treatment group, visit, and treatment-by-visit interaction as fixed effects, the baseline value of the response variable as a covariate, and subject as a random effect. Placebo is used as the reference group; Test type: Other; p = 0.3811, Mixed Effect Model Repeat Measurement
Statistical Analysis 2: Comparison: Placebo vs Leu Met Sil 1.0mg; [analysis description as in outcome 2, analysis 1]; Test type: Other; p = 0.8479, Mixed Effect Model Repeat Measurement

3. Secondary Outcome: Change in Circulating Cytokeratin 18 Fragments (M30)
Description: Change in Circulating Cytokeratin 18 Fragments (M30) from Baseline to Week 16 will be examined through standard blood chemistry
Time Frame: Baseline, Day 112
Population: For the Per-Protocol Population (N=70), the mean change (SD) in circulating cytokeratin 18 fragments (M30, U/L) from Baseline to week 16 was assessed
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Placebo | Leu Met Sil 0.5mg | Leu Met Sil 1.0mg
Number analyzed (Participants) | 22 | 24 | 24
U/L | 70.685 (306.3480) | 55.386 (273.1235) | 37.847 (222.6792)
Statistical Analysis 1: Comparison: Placebo vs Leu Met Sil 0.5mg; [analysis description as in outcome 2, analysis 1]; Test type: Other; p = 0.7742, Mixed effect Model Repeat Measurement
Statistical Analysis 2: Comparison: Placebo vs Leu Met Sil 1.0mg; [analysis description as in outcome 2, analysis 1]; Test type: Other; p = 0.6666, Mixed effect Model Repeat Measurement

4. Secondary Outcome: Change in Heamoglobin A1c (HbA1c)
Description: HbA1c will be examined through standard blood chemistry
Time Frame: Baseline, Day 112
Population: For the Per-Protocol Population (N=70), the mean change (SD) in HbA1c from Baseline to Week 16 was assessed.
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Placebo | Leu Met Sil 0.5mg | Leu Met Sil 1.0mg
Number analyzed (Participants) | 22 | 24 | 24
percentage | 0.07 (0.125) | -0.15 (0.287) | -0.11 (0.250)
Statistical Analysis 1: Comparison: Placebo vs Leu Met Sil 0.5mg; [analysis description as in outcome 2, analysis 1]; Test type: Other; p = 0.0020, MMRM
Statistical Analysis 2: Comparison: Placebo vs Leu Met Sil 1.0mg; [analysis description as in outcome 2, analysis 1]; Test type: Other; p = 0.0164, MMRM

5. Secondary Outcome: Change in Fasting Glucose
Description: Fasting glucose will be examined through standard fasting blood chemistry
Time Frame: Baseline, Day 112
Population: For the Per-Protocol Population (N=70), the mean change (SD) in fasting glucose from Baseline to Week 16 was assessed. The difference in the actual participants analyzed and per protocol population is due to missing or technically erroneous data.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | Leu Met Sil 0.5mg | Leu Met Sil 1.0mg
Number analyzed (Participants) | 22 | 23 | 23
mg/dL | 0.8 (10.66) | -2.7 (11.59) | -6.3 (9.13)
Statistical Analysis 1: Comparison: Placebo vs Leu Met Sil 0.5mg; [analysis description as in outcome 2, analysis 1]; Test type: Other; p = 0.4099, MMRM
Statistical Analysis 2: Comparison: Placebo vs Leu Met Sil 1.0mg; [analysis description as in outcome 2, analysis 1]; Test type: Other; p = 0.1455, MMRM

6. Secondary Outcome: Change in Insulin
Description: Insulin levels will be examined through standard blood chemistry
Time Frame: Baseline, Day 112
Population: For the Per-Protocol Population (N=70), the mean change (SD) in insulin from Baseline to Week 16 was assessed. The difference in the actual participants analyzed and per protocol population is due to missing or technically erroneous data.
Measure: Mean (Standard Deviation); unit: μIU/mL
Arm/Group | Placebo | Leu Met Sil 0.5mg | Leu Met Sil 1.0mg
Number analyzed (Participants) | 22 | 23 | 23
μIU/mL | -8.30 (24.38) | -6.60 (12.30) | -5.30 (15.84)
Statistical Analysis 1: Comparison: Placebo vs Leu Met Sil 0.5mg; [analysis description as in outcome 2, analysis 1]; Test type: Other; p = 0.2559, MMRM
Statistical Analysis 2: Comparison: Placebo vs Leu Met Sil 1.0mg; [analysis description as in outcome 2, analysis 1]; Test type: Other; p = 0.9776, MMRM

7. Secondary Outcome: Change in Blood Lipids (Cholesterol)
Description: Lipid levels such as cholesterol will be examined by standard blood chemistry
Time Frame: Baseline, Day 112
Population: For the Per-Protocol Population (N=70), the mean change (SD) in total cholesterol from Baseline to Week 16 was assessed.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | Leu Met Sil 0.5mg | Leu Met Sil 1.0mg
Number analyzed (Participants) | 22 | 24 | 24
mg/dL | -0.8 (27.56) | -20.5 (28.02) | -5.9 (37.98)
Statistical Analysis 1: Comparison: Placebo vs Leu Met Sil 0.5mg; [analysis description as in outcome 2, analysis 1]; Test type: Other; p = 0.2265, MMRM
Statistical Analysis 2: Comparison: Placebo vs Leu Met Sil 1.0mg; [analysis description as in outcome 2, analysis 1]; Test type: Other; p = 0.8366, MMRM

8. Secondary Outcome: Change in Blood Lipids (High Density Lipoprotein:HDL)
Description: Lipid levels such as HDL will be examined by standard blood chemistry
Time Frame: Baseline, Day 112
Population: For the Per-Protocol Population (N=70), the mean change (SD) in LDL from Baseline to Week 16 was assessed. The difference in the actual participants analyzed and per protocol population is because HDL could not be calculated for some participants.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | Leu Met Sil 0.5mg | Leu Met Sil 1.0mg
Number analyzed (Participants) | 21 | 22 | 21
mg/dL | -1.0 (23.81) | -13.3 (27.16) | 1.2 (42.27)
Statistical Analysis 1: Comparison: Placebo vs Leu Met Sil 0.5mg; [analysis description as in outcome 2, analysis 1]; Test type: Other; p = 0.3470, MMRM
Statistical Analysis 2: Comparison: Placebo vs Leu Met Sil 1.0mg; [analysis description as in outcome 2, analysis 1]; Test type: Other; p = 0.6221, MMRM

9. Secondary Outcome: Change in Low Density Lipoproteins (LDL)
Description: Lipid levels such as LDL will be examined by standard blood chemistry
Time Frame: Baseline, Day 112
Population: For the Per-Protocol Population (N=70), the mean change (SD) in LDL from Baseline to Week 16 was assessed. The difference in the actual participants analyzed and per protocol population is because LDL could not be calculated for some participants.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | Leu Met Sil 0.5mg | Leu Met Sil 1.0mg
Number analyzed (Participants) | 21 | 22 | 21
mg/dL | -1.0 (23.81) | -13.3 (27.16) | 1.2 (42.27)
Statistical Analysis 1: Comparison: Placebo vs Leu Met Sil 0.5mg; [analysis description as in outcome 2, analysis 1]; Test type: Other; p = 0.3470, MMRM
Statistical Analysis 2: Comparison: Placebo vs Leu Met Sil 1.0mg; [analysis description as in outcome 2, analysis 1]; Test type: Other; p = 0.6221, MMRM

10. Secondary Outcome: Change in Triglycerides
Description: Lipid levels such as triglycerides will be examined by standard blood chemistry
Time Frame: Baseline, Day 112
Population: Geometric mean values are presented since the data were skewed. Corresponding arithmetic mean changes from baseline for Treatments A, B and C in the Per Protocol Population were +54.9, -48.9 and -28.0 mg/dL respectively. This accounts for the p-value of p=0.0129 for Treatment B.
Measure: Geometric Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Leu Met Sil 0.5mg | Leu Met Sil 1.0mg
Number analyzed (Participants) | 22 | 24 | 24
mg/dL | 1.0 (0.06) | 0.8 (0.06) | 0.9 (0.06)
Statistical Analysis 1: Comparison: Placebo vs Leu Met Sil 0.5mg; [analysis description as in outcome 2, analysis 1]; Test type: Other; p = 0.0129, MMRM
Statistical Analysis 2: Comparison: Placebo vs Leu Met Sil 1.0mg; [analysis description as in outcome 2, analysis 1]; Test type: Other; p = 0.4316, MMRM

11. Secondary Outcome: Change in C-reactive Protein
Description: CRP levels will be examined by standard blood chemistry
Time Frame: Baseline, Day 112
Population: For the Per-Protocol Population (N=70), the geometric mean change (SE) in C-reactive protein from Baseline to Week 16 was assessed. The difference in the actual participants analyzed and per protocol population is due to missing or technically erroneous data.
Measure: Geometric Mean (Standard Error); unit: mg/L
Arm/Group | Placebo | Leu Met Sil 0.5mg | Leu Met Sil 1.0mg
Number analyzed (Participants) | 21 | 24 | 24
mg/L | 1.02 (0.129) | 1.27 (0.178) | 1.08 (0.170)
Statistical Analysis 1: Comparison: Placebo vs Leu Met Sil 0.5mg; Test type: Other — MMRM model: with treatment group, visit, and treatment-by-visit interaction as fixed effects, the baseline value of the response variable as a covariate, and subject as a random effect. Placebo is used as the reference group; p = 0.1946, MMRM
Statistical Analysis 2: Comparison: Placebo vs Leu Met Sil 1.0mg; [analysis description as in outcome 2, analysis 1]; Test type: Other; p = 0.4697, MMRM

12. Secondary Outcome: Change in Insulin Sensitivity (HOMA-IR)
Description: HOMA-IR levels will be examined by standard blood chemistry
Time Frame: Baseline, Day 112
Population: For the Per-Protocol Population (N=70), the change in geometric mean (SE) in HOMA-IR from Baseline to Week 16 was assessed. The difference in the actual participants analyzed and per protocol population is due to missing or technically erroneous data.
Measure: Geometric Mean (Standard Error); unit: mU/L
Arm/Group | Placebo | Leu Met Sil 0.5mg | Leu Met Sil 1.0mg
Number analyzed (Participants) | 20 | 22 | 22
mU/L | 0.89 (0.076) | 0.80 (0.078) | 0.85 (0.096)
Statistical Analysis 1: Comparison: Placebo vs Leu Met Sil 0.5mg; [analysis description as in outcome 2, analysis 1]; Test type: Other; p = 0.3474, MMRM
Statistical Analysis 2: Comparison: Placebo vs Leu Met Sil 1.0mg; [analysis description as in outcome 2, analysis 1]; Test type: Other; p = 0.8832, MMRM

ADVERSE EVENTS:
Time Frame: 112 days
Description: Treatment-Emergent Adverse Event (TEAE) is defined as an adverse event occurring on or after the first dose of randomized study medication, or existing prior to the time of and worsening after the time of the first dose of randomized study medication.
Arm/Group | Placebo | Leu Met Sil 0.5mg | Leu Met Sil 1.0mg
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/34 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/24 | 1/34 | 1/32
Other Adverse Events (participants affected / at risk) | 18/24 | 25/34 | 26/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=24) | Leu Met Sil 0.5mg (N=34) | Leu Met Sil 1.0mg (N=32)
Appendicitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastritis erosive (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=24) | Leu Met Sil 0.5mg (N=34) | Leu Met Sil 1.0mg (N=32)
Vision Blurred (Eye disorders) | 0 (0) | 2 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 3 (3) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 3 (3)
Blood triglycerides increase (Hepatobiliary disorders) | 0 (0) | 0 (0) | 2 (2)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1)
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 15 (15) | 12 (12)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 4 (4)
Dyspepsia (Gastrointestinal disorders) | 4 (4) | 3 (3) | 2 (2)
Fatigue (Social circumstances) | 1 (1) | 2 (2) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1) | 3 (3) | 4 (4)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Headache (General disorders) | 2 (2) | 5 (5) | 1 (1)
Nausea (General disorders) | 3 (3) | 6 (6) | 5 (5)
Type 2 Diabetes mellitus (Endocrine disorders) | 0 (0) | 1 (1) | 2 (2)
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 1 (1)
Vision blurred (Eye disorders) | 0 (0) | 2 (2) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 5 (5) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No